CLINICAL TRIAL: NCT06352281
Title: An Investigator-initiated Trial to Evaluate the Efficacy and Safety of CAR-T Cells Therapy in the Treatment of Chronic or Refractory Primary Immune Thrombocytopenia (ITP)
Brief Title: Efficacy and Safety of CAR-T Cells Therapy for Chronic or Refractory Primary Immune Thrombocytopenia (ITP)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: 920th Hospital of Joint Logistics Support Force of People's Liberation Army of China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KM-007
Record Dates: First submitted 2024-04-02; First posted 2024-04-08 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: ITP - Immune Thrombocytopenia
Keywords: CAR-T; Immune Thrombocytopenia (ITP)
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — Immunotherapy, Adoptive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CAR-T Cells Therapy (Experimental): Subjects who meet the enrollment conditions will receive intravenous infusion of CAR-T cells after lymphodepletion.
  Interventions: Biological: CAR-T cells

INTERVENTIONS:
Biological: CAR-T cells — CAR-T cells will be administered by vein. Before CAR-T infusion，patients will get a 3-5 days lymphodepletion therapy with fludarabine and cyclophosphamide.

SUMMARY:
It is a single-center, single-arm, open-labeled clinical trial to evaluate the efficacy and safety of CAR-T cells therapy for Chronic or Refractory Primary Immune Thrombocytopenia (ITP).

DETAILED DESCRIPTION:
This open label and single-arm study aims to evaluate the efficacy and safety of CAR-T cells therapy in patients with Chronic or Refractory Primary Immune Thrombocytopenia (ITP). After enrollment, a leukapheresis procedure will be performed to manufacture chimeric antigen receptor (CAR) modified T cells. Patients will get a 3-5 days lymphodepletion therapy with fludarabine and cyclophosphamide, then the CAR-T cells will be infused by vein. After infusion, subjects will be followed for safety and efficacy evaluation up to 12 weeks. For those with a durable remission 12 weeks after infusion, the follow-up will last for at least 12 months for disease control.

ELIGIBILITY:
Inclusion Criteria:

1. Willingness to complete the informed consent process and to comply with study procedures and visit schedule;
2. Men and women aged 8-75;
3. Participants diagnosed with chronic (>12 months duration) or refractory (a documented intolerance or insufficient response to the first and second line standard treatment of ITP) ITP;
4. The results of physical, instrumental, and laboratory examination of patients not suggest any disease which may cause thrombocytopenia other than ITP;
5. Platelet count <30 x 109 / L;
6. If the patient is taking corticosteroids, the treatment regimen/dose should be stable (at least 2 weeks prior to screening);
7. The results of physical, instrumental, and laboratory examination of patients should be within the normal range or deviations should be regarded by the researcher as clinically insignificant;
8. Willingness to use effective and reliable methods of contraception throughout the entire study period;

Exclusion Criteria:

1. All subjects with diseases which may cause secondary immune thrombocytopenia
2. Patients with preventive splenectomy;
3. Hemostatic disorders other than chronic thrombocytopenia;
4. Subject treated with drugs that affect platelet function (including but not limited to aspirin, clopidogrel and/or NSAIDs) or anti-coagulants for > 3 consecutive days within 2 weeks of the study start and until the end of the study;
5. History of platelet agglutination abnormality that prevents reliable measurement of platelet counts;
6. Concurrent malignant disease and/or history of cancer treatment with cytotoxic chemotherapy and/or radiotherapy;
7. Grade III-IV heart failure or myocardial infarction, cardiac angioplasty or stenting, unstable angina pectoris, or other clinically prominent heart disease within one year prior to enrollment;
8. History of thrombosis or presence of significant risk factors for thrombosis;
9. Persons with acute or exacerbation of chronic diseases of the gastrointestinal tract associated with the risk of bleeding, acute infectious diseases, pathologies of the respiratory system;
10. Any clinically significant hepatic impairment (increase of serum transaminase levels by more than 3 times the upper limit of normal);
11. Serum creatinine levels are more than two times higher than the upper limit of normal for a given age and sex;
12. Any other concomitant decompensated diseases or acute conditions, the presence of which, according to the researcher, may significantly affect the results of the study;
13. Human immunodeficiency virus (HIV) seropositivity, Hepatitis B surface antigen positive or hepatitis B core antibody positive and HBV-DNA positive, Patients with hepatitis C (HCV-RNA quantitative test results positive), Or the presence of other serious active viral or bacterial infections or uncontrolled systemic fungal infections;
14. Patients with severe history of allergy or allergic constitution;
15. Pregnancy and lactation;
16. History of mental illness and known alcohol/drug addiction;
17. Poor compliance due to physiological, family, social, geographical and other factors, unable to cooperate with the study protocol and follow-up plan;
18. Had undergone other clinical trials in the 4 weeks prior to participating in this trial;

Ages: 8 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Portion of patients with response (R) | At least 2 weeks after infusion
  platelet count>30x10^9/L and at least 2-fold increase of the baseline count, confirmed on at least 2 separate occasions at least 7 days apart, and absence of bleeding

SECONDARY OUTCOMES:
Portion of patients with complete response (CR) | At least 2 weeks after infusion
  platelet count>100x10^9/L, confirmed on at least 2 separate occasions at least 7 days apart, and absence of bleeding
Portion of patients with relapse | At least 2 weeks after infusion
  platelet count below 30x10^9/L or less than 2-fold increase of baseline platelet count or bleeding after treating effectively; platelet counts confirmed on at least 2 separate occasions approximately 1 day apart
Time (in days) from treatment start to response (R) | At least 2 weeks after infusion
  Time calculated from infusion to the day when the response (R) criteria are achieved
Time (in days) from treatment to complete response (CR) | At least 2 weeks after infusion
  Time calculated from infusion to the day when the complete response (CR) criteria are achieved
Duration (in days) of response (R) | At least 2 weeks after infusion
  Time calculated from the day when the response (R) criteria are achieved, to the day when loss of response (R) criteria is achieved
Incidence of adverse events(AE) after infusion | Up to 12 months after infusion
  The frequency, severity, and laboratory findings of all adverse events/serious adverse events are included. Description, time, classification, and outcome of AE events resulted from the investigational medical product, delivery method, or emergency measures will be recorded in the case report form.

CONTACTS AND LOCATIONS:
Overall Officials: Sanbin Wang, Doctor, Principal Investigator — 920th Hospital of Joint Logistics Support Force of People's Liberation Army of China
Locations (1):
- 920th Hospital of Joint Logistics Support Force of People's Liberation Army of China, Kunming, Yunnan, China